CLINICAL TRIAL: NCT06914973
Title: Evaluation of Corneal Epithelial Mapping in Diagnosis of Early Keratoconus by Anterior Segment Optical Coherence Tomography
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Refaat Nagib, residant doctor, Assiut University
Other Study IDs: mapping keratoconus OCT
Record Dates: First submitted 2025-03-25; First posted 2025-04-07 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group I: Control Group who intended to do LASIK (N=50)
- Group II: Keratoconus Group (N=50)
- Group III: Suspicious keratoconus by pentacam ( N=50)

SUMMARY:
The cornea, as the outermost refractive structure of the eye, plays a critical role in maintaining clear vision. Its transparency and structural integrity are essential for optimal visual function. Among the layers of the cornea, the corneal epithelium is of particular interest due to its dynamic nature and its ability to remodel in response to various physiological and pathological conditions. Accurate and repeatable measurement of corneal epithelial thickness (CET) is therefore crucial for diagnosing and managing corneal diseases, such as keratoconus, and for planning refractive surgeries Keratoconus, a progressive corneal ectatic disorder, is characterized by thinning and protrusion of the cornea, leading to irregular astigmatism and visual impairment. Early detection and monitoring of keratoconus rely heavily on precise corneal imaging, including CET mapping. While AS-OCT has shown promise in evaluating CET in both healthy and keratoconic eyes, the repeatability of these measurements must be thoroughly evaluated to ensure their clinical utility Early diagnosis with subsequent corneal crosslinking (CXL) can slow-down or stop keratoconus progression.9 Identifying subclinical keratoconus is extremely important in refractive surgery screening to avoid iatrogenic ectasia. Anterior and posterior corneal topography combined with total cornea thickness measurements and localisation of the thinnest area are the parameters used commonly for diagnosing and staging of corneal ectasias. Recently, epithelial thickness is also added as an additional parameter and is shown to be useful for both early diagnosis and grading of keratoconus Corneal imaging is an essential tool in modern eye care. Initially, the curvature of the anterior corneal surface constituted the ground for the estimation of corneal optical properties and diagnosis of ectatic disorders like keratoconus. Gradually the importance of the posterior corneal curvature as well as its thickness gained significance. In recent years, new imaging devices allowing fast and high-resolution imaging of the entire anterior segment, cornea included started to emerge. The main advantages of the new generation Anterior Segment Optical Coherence Tomography (AS-OCT) are their superior acquisition speed, improved optical resolution (axial and transversal), as well as scanning depth and field of view .

High-resolution imaging of the cornea with AS-OCT provides thickness measurements individually for epithelium and stroma individually. Measuring corneal epithelial thickness adds information that could be of value in early diagnosis, progression evaluation and maybe even for a more complete understanding of the pathophysiology of this disease. It has been shown that changes in the corneal epithelial thickness could be a sensitive tool for early keratoconus detection as well as for the assessment of the disease progression.

Precise measurements of the epithelial thickness are therefore important for keratoconus diagnosis and follow-up. AS-OCTs have high axial resolution and studies have shown that these instruments provide repeatable epithelial measurements both in central and peripheral cornea. With an additional lens (anterior segment module), posterior segments OCTs can also be used to measure corneal parameters including epithelial thickness1and previous studies have shown that these modules can also produce precise epithelial thickness measurements in healthy corneas and in keratoconus. There is only limited information on how the precision of epithelial measurements with the anterior module in posterior segment OCTs compares to the precision of epithelial measurements with AS-OCTs Aim of this study Detect early-stage keratoconus by identifying suitable epithelial thickness changes before topographic abnormalities appear .

- Provide higher accuracy compared to traditional topography by offering high-resolution cross-sectional imaging

ELIGIBILITY:
Inclusion Criteria:

* • Healthy participants with normal corneal topography and no ocular abnormalities intended to do LASIK.

  * Keratoconus patients with a confirmed diagnosis (based on corneal topography, tomography, and clinical signs).
  * Suspicious Keratoconus patients by pentacam.
  * Age ≥ 18 years.
  * Willingness to provide informed consent.

Exclusion Criteria:

* • History of corneal surgery or trauma.

  * Active ocular infection or inflammation.
  * Severe dry eye disease or other conditions affecting corneal epithelium.
  * Inability to cooperate with imaging procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients will be divided into three groups: healthy individuals , patients with keratoconus and suspicious keratoconus patient
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
epithelial thickness maps | baseline
  From the pachymetry map, we measured the central corneal thickness, and from the epithelial map, we measured central epithelial thickness, thickest location, thinnest location, and their distributionespecially in its subclinical or early stages.